CLINICAL TRIAL: NCT01328873
Title: A Prospective Assessment of the Diagnostic Utility of Emerging Laboratory Assessments Used in Conjunction With FOB in HSCT and Leukemia Patients With Acute Respiratory Symptoms and Pulmonary Infiltrates
Brief Title: FOB in HSCT and Leukemia Patients With Acute Respiratory Symptoms and Pulmonary Infiltrates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 909
Record Dates: First submitted 2011-03-01; First posted 2011-04-05 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Infiltrate New
Keywords: Pulmonary infiltrates; stem cell transplant; leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laboratory testing (Experimental): All patients will receive the lab testing on bronchoscopy specimens
  Interventions: Other: Microbiological analysis

INTERVENTIONS:
Other: Microbiological analysis — Bronchoalveolar lavage (BAL) with subsequent testing for pathogens

SUMMARY:
Pulmonary infiltrates frequently complicate the care of hematopoietic stem cell transplant (HSCT) and leukemia patients. Bronchoalveolar lavage (BAL) is frequently used to evaluate new pulmonary infiltrates in this population, however utility is limited by a historically low diagnostic yield for infection.

In an effort to improve diagnostic yields, this study will complete a Fiberoptic Bronchoscopy (FOB) within 8 hours of radiographic documentation of pulmonary infiltrates, prior to initiating new antibiotic therapy. To further improve detection of microbiological pathogens, the study will utilize PCR testing with rapid turnaround time to detect atypical pneumonia (M pneumoniae, C. Pneumonia, Legionella species, and respiratory viruses) and aspergillosis.

DETAILED DESCRIPTION:
Proper diagnosis and prompt treatment favorably impacts survival in the post transplant setting, but is often difficult and frequently results in inappropriate or late therapy. Low yields may be linked with empiric antibody therapy begun prior to the procedure, delayed time to procedure, procedure technique, the presence of graft versus host disease (GVHD), neutropenia, and diffuse infiltrates (as opposed to localized infiltrates or focal masses and nodules). One recent study found that early FOBs (less than or equal to 4 days between detection of pulmonary infiltrates and FOB) were 2.5 times more likely to establish a diagnosis of pneumonia compared to late examinations. Delaying this procedure(greater than 5 days between detection of pulmonary infiltrates and FOB) was associated with drug resistant organisms, polymicrobial infections, and worsened patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Autologous or allogeneic stem cell patients with new acute respiratory symptoms or pulmonary infiltrates
* leukemia patients with new acute respiratory symptoms or pulmonary infiltrates thought to be unrelated to disease

Exclusion Criteria:

* Patients unwilling to undergo FOB
* Patients unable to undergo FOB due to clinical status
* Patients unable to undergo FOB within 8 hours of radiographic report of pneumonia
* Patients unable to wait until completion of FOB to implement antibiotic changes
* Adults unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-03; Primary Completion 2015-10 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Kent Holland, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shannon VR, Andersson BS, Lei X, Champlin RE, Kontoyiannis DP. Utility of early versus late fiberoptic bronchoscopy in the evaluation of new pulmonary infiltrates following hematopoietic stem cell transplantation. Bone Marrow Transplant. 2010 Apr;45(4):647-55. doi: 10.1038/bmt.2009.203. Epub 2009 Aug 17. PMID 19684637
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Hardak E, Yigla M, Avivi I, Fruchter O, Sprecher H, Oren I. Impact of PCR-based diagnosis of invasive pulmonary aspergillosis on clinical outcome. Bone Marrow Transplant. 2009 Nov;44(9):595-9. doi: 10.1038/bmt.2009.65. Epub 2009 Mar 23. PMID 19308034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period - May 2011 - Sept 2015 Patients were identified in either the outpatient clinic or inpatient BMT/Leukemia unit
Pre-assignment Details: Patients were excluded only if they refused to participate or required antibiotic changes within the 7 days prior to being approached for the study. An additional 2 pateints were considered screen failures for this study and did not proceed.
Period: Overall Study
Arm/Group | Laboratory Testing
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Laboratory Testing
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants] — Patients were treated in an adult center. All patients were over the age of 18.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 36
    >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Positive Culture or Molecular Results After Brochoscopy
Description: To determine the diagnostic yield related to fiberoptic bronchoscopy (FOB) with bronchoalveolar lavage (BAL) in hematopoietic stem cell transplant (HSCT) and leukemia patients with acute respiratory symptoms and pulmonary infiltrates utilizing both current standard of care microbiology testing and emerging molecular genetic laboratory assessments.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | All Patients Will Receive Lab Testing on Bronchoscopy Specimen
Number analyzed (Participants) | 49
participants | 40

2. Secondary Outcome: Number of Patients With Positive CT Result
Description: To correlate specific types of pulmonary infiltrates (focal, multifocal, or diffuse interstitial or alveolar infiltrates) with microbiological findings. Patients were evaluated by changes on the CT and categorized as follows:
  1. Air space
  2. ground glass/reticular nodular
  3. nodular/cavitary
  4. single patchy infiltrate
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- Laboratory Testing: Patients were evaluated by changes on the CT and categorized as follows:
  1. Air space
  2. ground glass/reticular nodular
  3. nodular/cavitary
  4. single patchy infiltrate
  These were evaluated on CT scans and all units of measure are the same.
Arm/Group | Laboratory Testing
Number analyzed (Participants) | 49
participants | 49

3. Secondary Outcome: Number of Participants With Positive Bacterial Results by PCR
Description: To describe the microbiological findings in HSCT and leukemia patients with fever, respiratory symptoms, and pulmonary infiltrates
Time Frame: 24-48 hours
Measure: Number; unit: participants
Arm/Group | Laboratory Testing
Number analyzed (Participants) | 49
participants | 2

4. Secondary Outcome: Number of Patients With Positive Fungal Results by PCR
Description: as for outcome 3
Time Frame: 24-48 hours
Measure: Number; unit: participants
Arm/Group | Laboratory Testing
Number analyzed (Participants) | 49
participants | 4

5. Secondary Outcome: Number of Participants With Positive Viral Results by PCR
Description: as for outcome 3
Time Frame: 24-48 hours
Measure: Number; unit: participants
Arm/Group | Laboratory Testing
Number analyzed (Participants) | 49
participants | 48

6. Secondary Outcome: Number of Participants With Positive Myocbacteria Results by Culture
Description: as for outcome 3
Time Frame: 24-48 hours
Measure: Number; unit: participants
Arm/Group | Laboratory Testing
Number analyzed (Participants) | 49
participants | 2

ADVERSE EVENTS:
Arm/Group | Laboratory Testing
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications will need prior written consent from sponsor.